CLINICAL TRIAL: NCT00104195
Title: Decision-Making Processes and Brain Function in Anxiety-Disordered and Non-Anxious Youth
Brief Title: A Research Study of How Teens With and Without an Anxiety Disorder Make Decisions
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, F. Xavier Castellanos, Professor, NYU Langone Health
Other Study IDs: H11610
Record Dates: First submitted 2005-02-23; First posted 2005-02-24 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Anxiety Disorders; Separation Anxiety Disorder; Phobic Disorders
Keywords: Anxiety; Adolescence; Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Anxiety, Separation; Phobic Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this trial is to study how teens with and without an anxiety disorder make decisions.

This is a brain imaging study using functional magnetic resonance imaging (fMRI) in adolescents between the ages of 13 and 17.

DETAILED DESCRIPTION:
Preliminary analyses of behavioral data showed no group differences in response times during the decision-making games. However, behavioral ratings of certainty during the task showed differences between groups. Anxiety-disordered participants indicated lower levels of certainty during the most uncertain conditions of the task (p < .05). This difference was consistent with the study hypothesis. Within-subjects analyses of the decision-making tasks showed that subjects responded as expected. Reaction times (RT) during uncertain conditions of the HiLo-Game were significantly longer than during more certain conditions (p = .001). Diary Task RTs for rating ambiguous situations were significantly longer than ratings of unambiguous situations (p = .019). Preliminary Analyses showed a significant correlation between Intolerance of Uncertainty (IU) and RT during the Marble Task (r = -0.54, p < .05). Preliminary analysis also showed significant correlation between ratings of level of anxiety during the diary task and IU, IS, MASC and the child version of the SCARED. These preliminary results were not submitted for publication.

ELIGIBILITY:
Inclusion Criteria:

* Must meet diagnostic criteria for Generalized Anxiety Disorder, Separation Anxiety Disorder or Social Phobia, OR must be free of medical, psychiatric, neurologic conditions and learning disorders (healthy controls)
* Sufficient intelligence to understand the study and provide truly informed consent; will be determined by educational history

Exclusion Criteria:

* Having any major medical conditions that may interfere with interpretation of results or be associated with risk in an MRI environment (history of metal implants, or contraindications to MRI scanning for research purposes, including pregnancy)
* Current evidence of Autism, Major Depression, Substance Abuse, Obsessive Compulsive Disorder, Post-traumatic Stress Disorder, Panic Disorder, Tic Disorders, significant suicidality, lifetime history of psychosis or mania.
* Estimated Full-Scale IQ below 80
* Inability or unwillingness to remain still during scanning
* Inability or unwillingness to provide assent
* Absence of signed consent by parent or legal guardian
* Current history of sexual or physical abuse in the family, or past sexual or physical abuse if there is ongoing Department of Social Services (DSS) involvement

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Anxious and healthy adolescents
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2004-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Intolerance of Uncertainty | at time of assessment/enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- New York University's Child Study Center, New York, New York, United States